CLINICAL TRIAL: NCT06732843
Title: Does Recombinant FSH (rFSH, i.g. Gonal F®) as Compared to Human Menopausal Gonadotrophin (hMG) Affect Telomere Length of Cumulus Cells During Antral Follicle Growth and Impact Blastocyst Status?
Acronym: rFSH and hMG
Status: Recruiting | Type: Observational
Sponsor: ART Fertility Clinics LLC (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 2212-ABU-012-DN
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: OVARIAN STIMULATION; Telomere Length; Telomere Length, Mean Leukocyte
Keywords: recombinant human follicle-stimulating hormone (rFSH); uman-menopausal-gonadotropin (hMG; ocyte quality; embryo quality; blastocyst development; Menopur; GonalF; GnRH antagonist cycles; trophectoderm; cumulus cells

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Biospecimen Retention: Samples With DNA — Blood, cumulus cells and trophectoderm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Normo-ovarian response patients who undergo an IVF treatment including PGT-A: Patients will follow the stimulation protocol outlined below:
  Initial doses will be based on ovarian reserve parameters, with the starting dosage identical for both stimulation cycles (Gonal-F® or hMG):
  Dose adjustments may be made starting from day 6 Antagonist suppression will be fixed from day 5 onwards Final oocyte maturation will be triggered with a dual trigger: 2,500 IU urinary hCG and 0.3 mg Decapeptyl.

SUMMARY:
Gonal-F® (follitropin alfa) is a recombinant FSH without LH activity, while Menopur® contains both LH and hCG. The MEGASET trial compared Menopur® and Gonal-F® in GnRH antagonist cycles with SET, showing similar efficacy. A subsequent study (MEGASET-HR) in high responders found ongoing pregnancy rates of 35.5% for Menopur® and 30.7% for Gonal-F®, with a lower early pregnancy loss for Menopur® (14.5% vs 25.5%).

Telomere length (TL) in oocyte cumulus cells (CC) correlates with oocyte quality and embryo outcomes. This study aims to assess whether stimulation type (hMG vs. Gonal-F) affects TL in CC and subsequent blastocyst development. A randomized, open-label, cross-over study in normo-responders will analyze telomere length, embryo quality, and hormonal markers.

DETAILED DESCRIPTION:
Gonal-F® (follitropin alfa) is a recombinant human follicle-stimulating hormone (rFSH), without LH activity. Urine-derived, human-menopausal-gonadotropin contains LH and hCG. A highly purified hMG, HP-HMG, Menopur® has been compared with Gonal-F® in terms of ongoing pregnancy rate in the so called MEGASET trial ("Menopur in GnRH Antagonist Cycles with Single Embryo Transfer") and both showed to be effective in GnRH antagonist cycles with SET. Another non-inferiority study was initiated in high responders - MEGASET-HR-, comparing Menopur with Gonal-F. After fresh transfer, the ongoing pregnancy rate was similar between groups: 35.5% for Menopur versus 30.7% for Gonal-F, and non-inferiority was established. However, cumulative early pregnancy loss from fresh embryo transfer cycles (ET) and frozen embryo transfer cycles (FETs) in patients treated with HP-hMG was significantly lower as compared to rFSH (14.5% vs 25.5%).

Telomere length (TL) has been long proposed as oocyte quality marker and, recently, has been correlated with pregnancy outcomes. During folliculogenesis, granulosa cells undergo successive cell divisions which can result in telomeric shortening. Telomerase is the enzyme complex that binds the chromosome ends (telomeres) and maintains telomere length and integrity. An association has been shown between telomere length in cumulus cells (CC), oocyte competence and embryo quality. Hence, with the present study, the investigators aim to explore whether the stimulation treatment type (hMG versus Gonal-F) affects the telomere length of oocytes cumulus cells reflecting on subsequent blastocyst development, to help understanding the underlying differences between both gonadotropins.

To the investigators best knowledge, there are no studies evaluating TL in CC from the same patient exposed to two different stimulations. With the present, we intend to perform a randomized, open-label, cross-over study in a selected normo-responders patient population. Patients will be submitted to hormonal analysis, to analysis of telomere length of their oocyte cumulus cells and to analysis of quality markers of its respective embryos/blastocysts. This includes morphokinetics development, euploidy and mitochondria status evaluation of cultured blastocysts.

ELIGIBILITY:
Inclusion Criteria:

1. Maternal age 18 - 38 years
2. Patients requested PGT-A
3. BMI 18- 30kg/m2
4. Expected normoresponders
5. Fresh autologous ejaculate (≥5 mill/ml)
6. Sperm abstinence: 2-3 days
7. Normal female/male karyotype
8. Regular menstrual cycle length: 25-32 days
9. AFC of 5-10 in each ovary at the beginning of the stimulation
10. Trigger: dual trigger: 2.500 IU urinary hCG + 0.3 mg Decapeptyl. (13)
11. A wash-out period between 1 to 3 months; an inter-cycle variation of 10% in AFC, measured by the same physician, is accepted.
12. Couple agrees to perform two stimulations before continuing with embryo transfer

Exclusion Criteria:

* 1. Uterine abnormalities as diagnosed by ultrasound 2. Any hormonal or oral contraceptive pretreatment of 3 months preceding the treatment 3. Endometriosis according to American Fertility Society (AFS) ≥3 4. ≥ 2 miscarriages 5. Bologna criteria poor responders (14)

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Study Population: Normo-ovarian response patients who undergo an IVF treatment.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
In this study the investigators will investigate the telomere length of cumulus cells between two stimulation cycles, using different stimulation medication (rFSH versus hMG) within same patient/woman | 12 weeks
  In this study the investigators will investigate the telomere length of cumulus cells between two stimulation cycles, using different stimulation medication (rFSH versus hMG) within same patient/woman

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Lawrenz, PhD, Study Director — ART Fertility Clinics LLC
Locations (1):
- ART Fertility Clinics, Abu Dhabi, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yu TN, Cheng EH, Tsai HN, Lin PY, Chen CH, Huang CC, Lee TH, Lee MS. Assessment of Telomere Length and Mitochondrial DNA Copy Number in Granulosa Cells as Predictors of Aneuploidy Rate in Young Patients. J Clin Med. 2022 Mar 25;11(7):1824. doi: 10.3390/jcm11071824. PMID 35407431
- [Background] Gardner DK, Schoolcraft WB. Culture and transfer of human blastocysts. Curr Opin Obstet Gynecol. 1999 Jun;11(3):307-11. doi: 10.1097/00001703-199906000-00013. PMID 10369209
- [Background] Younis JS, Ben-Ami M, Ben-Shlomo I. The Bologna criteria for poor ovarian response: a contemporary critical appraisal. J Ovarian Res. 2015 Nov 17;8:76. doi: 10.1186/s13048-015-0204-9. PMID 26577149
- [Background] Haas J, Bassil R, Samara N, Zilberberg E, Mehta C, Orvieto R, Casper RF. GnRH agonist and hCG (dual trigger) versus hCG trigger for final follicular maturation: a double-blinded, randomized controlled study. Hum Reprod. 2020 Jul 1;35(7):1648-1654. doi: 10.1093/humrep/deaa107. PMID 32563188
- [Background] Butts S, Riethman H, Ratcliffe S, Shaunik A, Coutifaris C, Barnhart K. Correlation of telomere length and telomerase activity with occult ovarian insufficiency. J Clin Endocrinol Metab. 2009 Dec;94(12):4835-43. doi: 10.1210/jc.2008-2269. Epub 2009 Oct 28. PMID 19864453
- [Background] Liu JP, Li H. Telomerase in the ovary. Reproduction. 2010 Aug;140(2):215-22. doi: 10.1530/REP-10-0008. Epub 2010 Jun 18. PMID 20562297
- [Background] Fu D, Collins K. Purification of human telomerase complexes identifies factors involved in telomerase biogenesis and telomere length regulation. Mol Cell. 2007 Dec 14;28(5):773-85. doi: 10.1016/j.molcel.2007.09.023. PMID 18082603
- [Background] Riethman H, Ambrosini A, Paul S. Human subtelomere structure and variation. Chromosome Res. 2005;13(5):505-15. doi: 10.1007/s10577-005-0998-1. PMID 16132815
- [Background] Vasilopoulos E, Fragkiadaki P, Kalliora C, Fragou D, Docea AO, Vakonaki E, Tsoukalas D, Calina D, Buga AM, Georgiadis G, Mamoulakis C, Makrigiannakis A, Spandidos DA, Tsatsakis A. The association of female and male infertility with telomere length (Review). Int J Mol Med. 2019 Aug;44(2):375-389. doi: 10.3892/ijmm.2019.4225. Epub 2019 May 31. PMID 31173155
- [Background] Cheng EH, Chen SU, Lee TH, Pai YP, Huang LS, Huang CC, Lee MS. Evaluation of telomere length in cumulus cells as a potential biomarker of oocyte and embryo quality. Hum Reprod. 2013 Apr;28(4):929-36. doi: 10.1093/humrep/det004. Epub 2013 Feb 1. PMID 23377770
- [Background] Kosebent EG, Uysal F, Ozturk S. Telomere length and telomerase activity during folliculogenesis in mammals. J Reprod Dev. 2018 Dec 14;64(6):477-484. doi: 10.1262/jrd.2018-076. Epub 2018 Sep 28. PMID 30270279
- [Background] 5. J. Michaeli, K. Rotshenker Olshinka, N. Srebnik, R. Smoom, N. Serruya, S. Yanai, O. Michaeli, T. Eldar-Geva, Y. Tzfati. Oral communication in ESHRE 2020 preselected for an award: The telomere link between extended fertility and longevity.
- [Background] Witz CA, Daftary GS, Doody KJ, Park JK, Seifu Y, Yankov VI, Heiser PW; Menopur in GnRH Antagonist Cycles with Single Embryo Transfer - High Responder (MEGASET-HR) Trial Group. Randomized, assessor-blinded trial comparing highly purified human menotropin and recombinant follicle-stimulating hormone in high responders undergoing intracytoplasmic sperm injection. Fertil Steril. 2020 Aug;114(2):321-330. doi: 10.1016/j.fertnstert.2020.03.029. Epub 2020 May 13. PMID 32416978
- [Background] Devroey P, Pellicer A, Nyboe Andersen A, Arce JC; Menopur in GnRH Antagonist Cycles with Single Embryo Transfer Trial Group. A randomized assessor-blind trial comparing highly purified hMG and recombinant FSH in a GnRH antagonist cycle with compulsory single-blastocyst transfer. Fertil Steril. 2012 Mar;97(3):561-71. doi: 10.1016/j.fertnstert.2011.12.016. Epub 2012 Jan 13. PMID 22244781
- [Background] van Wely M, Kwan I, Burt AL, Thomas J, Vail A, Van der Veen F, Al-Inany HG. Recombinant versus urinary gonadotrophin for ovarian stimulation in assisted reproductive technology cycles. Cochrane Database Syst Rev. 2011 Feb 16;2011(2):CD005354. doi: 10.1002/14651858.CD005354.pub2. PMID 21328276
- [Background] Fatemi HM. Assessment of the luteal phase in stimulated and substituted cycles. Facts Views Vis Obgyn. 2009;1(1):30-46. No abstract available. PMID 25478069